CLINICAL TRIAL: NCT02103530
Title: Early Response Assessment of Induction Chemotherapy in Acute Myeloid Leukemia Patients Using F-18 FLT PET/CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Woo Hee Choi, MD, Clinical assistant professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VC13MISI0184
Record Dates: First submitted 2014-02-03; First posted 2014-04-04 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLT PET/CT (Experimental): Patients who had FLT PET/CT
  Interventions: Other: FLT PET/CT

INTERVENTIONS:
Other: FLT PET/CT — All PET/CT scans were performed using a hybrid PET/CT scanner (Gemini TF 64 with Astonish TF, Philips). F-18 FLT (2.96 MBq/kg) in 2-5 mL of normal saline was injected intravenously. One hour after FLT injection, CT began at the vertex and progressed to the upper thigh (120 kVp, 100 mA and 4 mm slice thickness). PET emission data were acquired immediately for 1 min at each bed position followed. The CT data were used for attenuation correction. Images were reconstructed using a standard ordered-subset expectation maximization algorithm with 3 iterations and 33 subsets.

SUMMARY:
The purpose of this study is to investigate whether F-18 FLT PET/CT is useful in early response assessment of induction chemotherapy in acute myeloid leukemia patients.

DETAILED DESCRIPTION:
Assessment of treatment response in AML is very important to determine the next treatment. Standard treatment of AML begins with induction chemotherapy. NCCN guideline recommend to assess the treatment response via bone marrow examination approximately 7-10 days after completion of induction chemotherapy. However, the possibility of sampling error and risks of infection and bleeding are the limitation of bone marrow biopsy.

F-18 fluorodeoxythymidine (FLT) is a radiopharmaceutical for PET, reflecting the proliferation of the cell. F-18 FLT is trapped after phosphorylation by thymidine kinase1, whose expression is increased in replicating cells. There have been several studies that reported F-18 FLT PET could measure health and proliferation of the bone marrow.

The aim of this study is to evaluate if F-18 FLT PET/CT is suitable for early response assessment of induction chemotherapy in acute myeloid leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

* acute myeloid leukemia
* must receive induction chemotherapy
* 19 years old and over

Exclusion Criteria:

* no standard therapy
* pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Value of FLT PET/CT in early response assessment of induction chemotherapy in acute myeloid leukemia | 4-6 wks after completion of induction chemotherapy
  Correlation between the FLT PET/CT findings on day 8-12 after start of treatment with the result of bone marrow biopsy which is done 4-6 wks after completion of induction chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Woo Hee Choi, MD, Principal Investigator — St. Vincent's Hospital, The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyenggi-do, South Korea